CLINICAL TRIAL: NCT05809193
Title: Investigation of the Effects of Family-Focused Therapy in the Early Period of Bipolar Disorder and Psychotic Disorder
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Dokuz Eylul University (Other)
Responsible Party: Principal Investigator, Tevhide Ekin Sut, M.D., Department of Child and Adolescent Psychiatry, Dokuz Eylul University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2022/11-07
Record Dates: First submitted 2023-03-27; First posted 2023-04-12 (Actual); Last update posted 2024-06-11 (Actual); Status verified 2024-06

CONDITIONS: Mental Disorder in Adolescence; Bipolar Disorder; Psychosis; Family Relations
Keywords: family focused therapy; bipolar disorder; psychotic disorder; child; adolescent; early intervention
MeSH Terms: conditions — Bipolar Disorder; Psychotic Disorders

STUDY DESIGN:
Intervention Model Description: It is aimed to examine the effects of family-focused therapy, which will be applied in the early period to individuals who have been diagnosed with bipolar disorder and psychotic disorder and who have achieved remission, and their families. It will be carried out using the guide "Family-Focused Therapy for High-Risk Adolescents and Young Adults for Bipolar Disorder or Psychosis" revised by Miklowitz et al. in 2018. In terms of practical application, the sessions will be psychoeducational sessions that will be held in groups of 3 sessions, 3 sessions with the youth and the family. communication skills sessions to be held individually and 3 sessions as problem solving skills sessions to be held individually with the youth and family will be completed in 9 sessions. Sessions will be held once a week and all sessions will be completed in 9 weeks.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Family-Focused Therapy (Experimental): Bipolar Disorder and Psychotic Disorder
  Interventions: Behavioral: Family-Focused Therapy

INTERVENTIONS:
Behavioral: Family-Focused Therapy — After the patient and family are informed, they are included in the therapy group on a voluntary basis. After evaluation by independent evaluators, therapy sessions are started by therapists.
  Session 1: Goal Setting, Treatment Overview, Symptoms, Vulnerability Stress Model Session 2: Stress and Coping Skills, Regulation of sleep habits, Relaxation exercises Session 3: Optimizing Family Support; Prevention Plan, Medication adherence Session 4: Overview of Communication Skills; Expressing Positive Feelings, Active Listening Session 5: Making Positive Requests for Change, Communication Clarity Session 6: Expressing Negative Feelings Session 7: Introduction to Problem Solving Skills Session 8 and 9: Problem Solving Skills, Termination of Treatment The same psychometric assessment will be repeated before and after FFT. Intra-group comparisons will be made. Also study groups will be compared using time by group interactions to investigate the differences in therapy response.

SUMMARY:
Family-focused therapy (FFT) is a comprehensive therapy approach applied to individuals and their families. In the present study, the researchers aimed to investigate the effects of family-focused therapy (FFT) in the early stages of psychotic disorder and bipolar disorder, regarding the psychiatric symptomatology, family communication skills, coping capacities, family burden and quality of life. A total of 34 young people diagnosed with bipolar disorder (BD) and 17 psychotic disorders (PD) will be included in the study.

DETAILED DESCRIPTION:
In this study, the researcher's primary goal is to investigate the effects of family-focused therapy sessions on young people aged between 15 and 21. Subjects were referred to an early intervention center for psychotic and bipolar disorders. The target population of the study consists of the patients in remission after the episode of the illness.

Therapy sessions will be conducted in line with the manual for "Family Focused Therapy for High-Risk Adolescents and Young Adults for Bipolar Disorder or Psychosis" revised by Miklowitz et al. in 2018. FFT will be completed in nine sessions. The first module of the program consists of three sessions, which consists of group psychoeducation for the patients and families. The second and third modules also include three sessions in each to teach communication skills and problem-solving skills in individual therapy sessions including patients and their families. Sessions will be held once a week and completed in nine weeks.

Within the scope of this program, non-therapist clinicians will evaluate the participants' symptoms, psychosocial functioning, insight, and treatment compliance before and after the therapy sessions.

There are only a few previous studies investigating the effects of family therapy in early stages of bipolar disorder and psychotic disorder. According to the literature, no prior study compares the effects of FFT between BD and PD populations. This study is important in terms of developing effective strategies for management of psychosocial difficulties in early phases of BD and PDs.

ELIGIBILITY:
Inclusion Criteria:

* Not be in an active phase of the illness
* Able to comply with the interviews
* The total score of the Hamilton Depression Rating Scale ≤ 21 points.
* The total score of the Young Mania Rating Scale ≤ 14 points.
* At least one family member with the capacity to read and write in Turkish

Exclusion Criteria:

* Neurological disorders and serious physical disease that affect cognitive functions
* The symptoms due to substance use or a medical illness
* Autism Spectrum Disorder
* Comorbid alcohol and substance abuse (except nicotine)
* Co-morbid psychiatric disorders except disruptive behavior disorders and anxiety disorders

Ages: 15 Years to 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 20 (Actual)
Dates: Start 2022-04-01 (Actual); Primary Completion 2023-10-01 (Actual); Study Completion 2023-12-31 (Actual)

PRIMARY OUTCOMES:
The change from baseline to follow-up in Hamilton Depression Rating Scale (HDRS) scores | at baseline and at week 9
  by independent clinician/ to the patient - HDRS is a clinician-administered scale that measures the severity of depression. It contains 17 questions scored between 0-4. The total score of the scale ranges from 0 to 51. Cut-off points were determined as <7 normal, 8-13 mild, 14-18 moderate, 19-22 severe and >23 very severe.
The change from baseline in Young Mania Rating Scale score | at baseline and at week 9
  by independent clinician/ to the patient - The Young Mania Rating Scale (YMRS) is a likert-type scale developed to measure the severity of manic symptoms. 7 of 11 items are graded in the range of 0-4, and the other 4 items are graded in the range of 0-8 points. Therapy sessions will be started if the Young Mania Rating Scale total score is ≤ 14 points. In addition, measurements will be repeated at the end of therapy.
The change from baseline in Scale for the Assessment of Positive Symptoms (SAPS) | at baseline and at week 9
  by independent clinician/ to the patient - This scale aims to measure severity of positive symptoms in schizophrenia. It includes a total of 34 items in 4 subscales: hallucinations, delusions, bizarre behavior and positive formal thought disorder. Measurements will be made at the beginning and the difference will be examined by repeating at the end of the sessions.
The change from baseline in Brief Negative Symptom Scale (BNSS) | at baseline and at week 9
  by independent clinician/ to the patient - BNSS consists of 13 items and has six subscales: anhedonia, stress, asociality, avolition, blunt affectivity, and alogia. The total score of the scale, which can range from 0 to 78, is obtained by summing the scores of 13 items. Measurements will be made at the beginning and the difference will be examined by repeating at the end of the sessions.
The change from Personal and Social Performance Scale (PSP) scores | at baseline and at week 9
  by independent clinician/ to the patient - The scale evaluates personal and social performance in 4 sub-dimensions; Socially useful activities, personal and social relationships, self-care, irritating and aggressive behavior. 6-point Likert-type rating (1=absent - 6=very severe) was used.
The change from Scale of Unawareness of Mental Disorder (SUMD) scores | at baseline and at week 9
  by independent clinician/ to the patient - SUMD was developed by Amador et al in 1993 to evaluate insight in psychiatric disorders. The Turkish reliability of this scale was determined by Bora E et al. (Bora et al. 2006). The scale is scored between 1-5 points and consists of 3 general items: being aware of mental disorders, being aware of the effects of drugs, and being aware of the social consequences of the disorder. High scores represent poor insight.

SECONDARY OUTCOMES:
Coping Strategies Scale Brief Form (Brief COPE) | at baseline and at week 9
  self report / to the patient - The Coping Strategies Short Form is the short form of the Coping Strategies (COPE) scale developed by Carver, Scheier, and Weintraub (1989), which measures people's different behaviors against stress, developed by Carver (1997). Coping Strategies Short Form consists of 14 subscales. It will be given at the beginning and at the end of the therapy sessions and the difference will be evaluated.
Shortened Level of Expressed Emotion Scale | at baseline and at week 9
  self report / to the patient - The scale developed by Nelis et al. consists of 33 items measuring the perceived emotional expression of the most influential person in the participant's life in the last three months. The three subscales of the scale are lack of emotional support, irritability and intrusiveness. It will be given at the beginning and at the end of the therapy sessions and the difference will be evaluated.
World Health Organization Quality of Life Assessment (WHOQOL) | at baseline and at week 9
  self report / to the patient and parent - The WHOQOL-BREF scale consists of a total of 26 questions, two questions about the general health, and 4 areas: physical health, psychological health, social relationships and environment. It will be given at the beginning and at the end of the therapy sessions and the difference will be evaluated.
Mc Master Family Assessment Device | at baseline and at week 9
  self report / to the patient and parent - The scale, which consists of seven subscales called Problem Solving, Communication, Roles, Affective Responsiveness, Affective Involvement, Behavior Control, and General Functioning, consists of 60 items. The scale is scored over four options varying between one and four points. Theoretically, two scores were accepted as a score distinguishing healthy and unhealthy functions. It can be applied to all family members over the age of twelve and to the subject himself to evaluate family functions. It will be given at the beginning and at the end of the therapy sessions and the difference will be evaluated.
Beck's Depression Inventory | at baseline and at week 9
  self report / to parent - It is a widely used self-report scale developed by Beck in 1961. The Beck's Depression Inventory consists of 21 items related to depressive symptoms such as pessimism, sense of failure, dissatisfaction, feelings of guilt, restlessness, fatigue, decreased appetite, indecision, sleep disturbance, and social withdrawal. Each item gets a score between 0 and 3. The highest possible score is 63.
Zarit Burden Interview | at baseline and at week 9
  self report / to parent - The scale, which can be filled in by the caregivers themselves or by the researcher, consists of 22 statements that determine the effect of caregiving on the individual's life. The scale has a Likert-type rating ranging from 0 to 4 as never, rarely, sometimes, often, or almost always.

CONTACTS AND LOCATIONS:
Overall Officials: Neslihan Inal, M.D., Study Director — Dokuz Eylul University Department of Child and Adolescent Psychiatry; Emre Bora, M.D., Study Director — Dokuz Eylul University Department of Psychiatry
Locations (1):
- Dokuz Eylül University, Izmir, Balcova, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No